CLINICAL TRIAL: NCT00780650
Title: Mechanisms of Hypoglycemia Associated Autonomic Dysfunction, Q4-Atomoxetine
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Stephen N. Davis, MBBS, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HP-00044873
Record Dates: First submitted 2008-10-24; First posted 2008-10-27 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Atomoxetine
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atomoxetine — 80 mg oral dose, once per day for 6 weeks
  Other Names: Strattera
  Arms: 1
Drug: Placebo — 80 mg dose once per day for 6 weeks
  Arms: 2

SUMMARY:
This study is aimed at determining if the drug Atomoxetine (Strattera-used to treat Attention Deficit Hyperactivity Disorder(ADHD) has effects on the body's ability to defend itself against low blood sugar.

DETAILED DESCRIPTION:
The purpose of this study is to see if the drug atomoxetine (Strattera) has effects on the body's ability to defend itself against low blood sugar. Normally, when blood sugar levels drop below normal, the body creates a series of responses, which increase the sugar inside the body to bring blood sugar levels back to normal. The hormone epinephrine is a key defense against low blood sugar in people with diabetes. Atomoxetine has been shown to increase this hormone level. Thus, any approaches to increase levels of this key defense during low blood sugar may have great value.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals aged 18-50 years
* Type 1 Diabetes individuals aged 18-50 years
* BMI <40 kg/m2
* Females of childbearing potential with negative urine pregnancy test
* Volunteers over 40 years of age, a cardiac stress test with no clinically significant conduction or ischemic changes

Exclusion Criteria:

The following groups of subjects will be excluded from the study:

* Pregnant women
* Subjects unable to give voluntary informed consent
* Subjects on anticoagulant drugs or with known bleeding diatheses
* Subjects with uncontrolled hypertension, heart disease, cerebrovascular incidents
* Subjects taking MAOIs
* Subjects with narrow angle glaucoma
* Subjects with diagnosed psychiatric disorders
* Subjects with allergy to atomoxetine, heparin, or lidocaine

Physical Exam Exclusion Criteria:

* Uncontrolled severe hypertension (i.e., blood pressure greater than 150/95)
* Clinically significant Cardiac Abnormalities (e.g. Heart Failure, Arrhythmias, ischemic tachycardia, S-T segment deviations, etc.) from history or from cardiac stress testing in subjects > 40 years old.
* Pneumonia
* Hepatic Failure/Jaundice
* Renal Failure
* Acute Cerebrovascular/ Neurological deficit
* Fever greater than 38.0 C

Screening Laboratory Tests Exclusion Criteria Blood values as defined in protocol

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2009-05; Primary Completion 2018-08-21 (Actual); Study Completion 2018-08-21 (Actual)

PRIMARY OUTCOMES:
Change in level of catecholamines in blood from baseline | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephen N. Davis, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Univerisity of Maryland, Baltimore, Baltimore, Maryland, United States